CLINICAL TRIAL: NCT05001243
Title: Comparison of Pilocarpine, Brimonidine, Oxymetazoline, Hialuronic Acid, Bromfenac Ophthalmic Compound With Pilocarpine and Brimonidine to Improve Uncorrected Visual Acuity in Healthy Presbyopic Individuals
Brief Title: Comparison of a Compound With Pilocarpine and Brimonidine to Improve Near Vision in Healthy Presbyopic Patients
Acronym: PBOHB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Optall Vision (Other)
Responsible Party: Principal Investigator, Cesar Alejandro Sanchez Galeana, Principal Investigator, Optall Vision
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBOCP3
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Brimonidine Tartrate; Oxymetazoline; Hyaluronic Acid; bromfenac; Pilocarpine; sepharose-4B-polyisoluminol

STUDY DESIGN:
Intervention Model Description: Single Group Assignment To determine safety and efficacy of a Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic Acid, Bromfenac compound compared to Brimonidine and Pilocarpine to improve near uncorrected vision in healthy presbyopic patients
Who Masked: Participant, Care Provider
Masking Description: While in office the care provider took a number out of a closed container. Number 1 was designated for the Brimonidine, Number 2 was designated for the PBOHB compound, Number 3 was designated for de Pilocarpine compound
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental PBOHB (Experimental): Pilocarpine, brimonidine, Oxymetazoline combined with Hyaluronic Acid and Bromfenac combined in an ophthalmic solution to be randomly instilled in one eye.
  Interventions: Drug: Pilocarpine Hydrochloride; Drug: Brimonidine Tartrate
- Pilocarpine 5 mgs (Active Comparator): Pilocarpine was instilled in the other oye.
  Interventions: Drug: Compound Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic acid, Bromfenac
- Brimonidine 0.5 mgs (Active Comparator): Brimonidine was instilled in the other eye.
  Interventions: Drug: Compound Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic acid, Bromfenac

INTERVENTIONS:
Drug: Compound Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic acid, Bromfenac — PBOHB to improve uncorrected near vision in healthy presbyopic patients
  Other Names: PBOHB
  Arms: Brimonidine 0.5 mgs; Pilocarpine 5 mgs
Drug: Pilocarpine Hydrochloride — Apply in the fellow eye
  Other Names: Pil
  Arms: Experimental PBOHB
Drug: Brimonidine Tartrate — Apply in the fellow eye
  Other Names: Brimonidine
  Arms: Experimental PBOHB

SUMMARY:
Safety and Efficacy of Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic acid, Bromfenac (PBOHB) ophthalmic compound compared to Pilocarpine and Brimonidine to improve uncorrected near vision in healthy presbyopic patients one hour after instillation.

DETAILED DESCRIPTION:
To determine the safety and efficacy of a novel pharmacological compound of Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic acid, Bromfenac (PBOHB) to improve uncorrected near vision in healthy presbyopic patients compared to Pilocarpine and Brimonidine one hour after binocular instillation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Presbyopic
* 40 - 59 years

Exclusion Criteria:

* Diabetics
* Previous eye surgery
* Previous eye disease
* > 0.50 myopia
* > 1.5 hyperopia or astigmatism

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
Number of eyes improving 3 lines or more near visual acuity | 1 hour
  Eyes instilled with PBOHB
Eyes improving 3 lines or more near visual acuity | 1 hour
  Eyes instilled with Pilocarpine
Eyes improving 3 lines or more near VA | 1 hour
  Eyes instilled with Brimonidine

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Alejandro S Galeana, MD, Principal Investigator — Optall Vision
Locations (1):
- Optall Vision, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No